CLINICAL TRIAL: NCT05528263
Title: Preventing Chemotherapy-Induced Peripheral Neuropathy With Acupuncture, A Randomized Controlled Trial (PACT Trial)
Brief Title: Preventing Chemotherapy-Induced Peripheral Neuropathy With Acupuncture (PACT Trial)
Acronym: PACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The Comprehensive and Integrative Medicine Institute of South Korea (Other)
Responsible Party: Principal Investigator, Weidong Lu, MB, MPH, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-269
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Acupuncture; Early-stage Breast Cancer; Chemotherapy-induced Peripheral Neuropathy; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: Acupuncture; Early-stage Breast Cancer; Chemotherapy-induced Peripheral Neuropathy; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acupuncture (Experimental): * Breast cancer patients will be recruited who are scheduled to receive taxane-based chemotherapy (with or without anti-HER2 therapy) and who have no neuropathic symptoms at baseline.
    40 participants will be randomized into the acupuncture Arm:
  * The acupuncture arm will receive a standardized acupuncture protocol 1-2 times a week for 12 weeks (a total of 14 sessions).
  Interventions: Device: Acupuncture
- Nature scenery videos with relaxation exercise (Active Comparator): * Breast cancer patients will be recruited who are scheduled to receive taxane-based chemotherapy (with or without anti-HER2 therapy) and who have no neuropathic symptoms at baseline.
    40 Participants will be randomized into the Control Arm:
  * The control arm will receive and watch videos with nature scenery with a relaxation exercise guide 1-2 times a week for 12 weeks (a total of 14 sessions)
  Interventions: Other: Nature scenery with a relaxation exercise

INTERVENTIONS:
Device: Acupuncture — Standardized acupuncture protocol 1-2 times a week for 12 weeks (a total of 14 sessions).
  Arms: Acupuncture
Other: Nature scenery with a relaxation exercise — Watch nature scenery videos with a relaxation exercise guide 1-2 times a week for 12 weeks (a total of 14 sessions)
  Arms: Nature scenery videos with relaxation exercise

SUMMARY:
This research is being done to determine whether acupuncture can help prevent or lessen chemotherapy-induced peripheral neuropathy (CIPN), a side effect of some kinds of chemotherapy that causes pain, numbness, tingling, swelling, or muscle weakness mostly in the hands or feet.

This research will also help determine whether acupuncture can improve quality of life in patients receiving taxane-based chemotherapy for the treatment of breast cancer.

The names of the study activities involved in this study are/is:

* Acupuncture treatments for participants in the Acupuncture Group
* Nature videos with a relaxation exercise for participants in the Relaxation/ Exercise Group

The Comprehensive and Integrative Medicine Institute (CIMI) of South Korea is supporting this research study by providing funding.

DETAILED DESCRIPTION:
This study randomly assigns patients with breast cancer who are starting a chemotherapy program that includes a Taxane to one of two groups:

* The Acupuncture Group will receive acupuncture treatments for 12 weeks during chemotherapy treatment.
* The Relaxation Exercise Group will receive a program of weekly videos accompanied by a relaxation exercise. Both programs will last 12 weeks.

Participants will be asked to complete questionnaire 12 weeks after the completion of the acupuncture or relaxation exercise program, so participants be on this research study for up to 24 weeks (6 months).

It is expected that about 80 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically proven stage I-III breast cancer, without evidence of distant metastasis
* Scheduled to receive adjuvant or neoadjuvant taxane-based chemotherapy (with or without HER-2 directed therapy or with or without immunotherapy). Patient must enroll before the second infusion of a taxane.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Signed informed consent

Exclusion Criteria:

* Previous receipt of CIPN-inducing chemotherapy agents (1 prior dose of a taxane is allowed).
* Unstable cardiac disease or myocardial infarction within 6 months prior to study entry
* Wearing a pacemaker or implantable cardioverter-defibrillator
* Uncontrolled seizure disorder
* History of pre-existing peripheral neuropathy
* Use of acupuncture within the 3 months prior to study enrollment
* Self-report of any CIPN symptoms via staff-administered PRO-CTCAE CIPN, defined as either:

  * Report of "mild", "moderate", "severe", "very severe" on the Severity Item on PRO-CTCAE CIPN assessment
  * Report of "a little bit", "somewhat", "quite a bit", "very much" on the Interfere Item on PRO-CTCAE CIPN assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in severity of CIPN, defined by mean change in EORTC QLQ-CIPN20 sensory score | baseline to 12 weeks
  The primary endpoint is the change in severity of CIPN, defined as the average change from baseline (12-week to baseline) in the EORTC Quality of Life - Chemotherapy Induced Neuropathy 20 (QLQ-CIPN20) sensory subscale score (9 items). Using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), individuals indicate the degree to which they have experienced sensory, motor, and autonomic symptoms during the past week. A higher score means greater severity of CIPN. The total and three domain scores are calculated and linearly transformed into 0-100 scales according to the scoring manual. A score of 100 indicates the worst CIPN symptom.

SECONDARY OUTCOMES:
Incidence of CIPN between intervention arms - AOCIPN | baseline to week 12
  AOCIPN is defined as an increase of 2.5 points or larger in the QLQ-CIPN 20 sensory score at any time point relative to baseline or reported "mild" or "a little bit" or higher in PRO-CTCAE CIPN "Severity" and "Interference" items during the study intervention period (baseline to week 12).
Incidence of CIPN between intervention arms - G2CIPN | baseline to 12 Weeks
  G2CIPN is defined a 20-point or greater increase from baseline at any time point in QLQ-CIPN20 total score or grade-2 in PRO-CTCAE CIPN, which is defined as reporting the severity of numbness and/or tingling AND interference of with daily activities ≥ 1 (mild/ a little bit) during the study period at any time point.
Relative dose intensity (RDI) | baseline to week 24
  Received or relative dose intensity (RDI) refers to the amount and timing of chemotherapy actually delivered versus the expected dose and schedule. The relative dose intensity (RDI) will be calculated for each participant and compared between treatment arms using two-sample t-tests or Wilcoxon rank-sum tests, depending upon normality of the data.
Maximum CIPN score | pre-treatment, and at weeks 3, 6, 9, and 12 during the intervention up to 12 weeks
  Maximum CIPN score will be assessed through the EORTC Quality of Life - Chemotherapy Induced Neuropathy 20 (QLQ-CIPN20) sensory subscale score (9 items). Using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), individuals indicate the degree to which they have experienced sensory, motor, and autonomic symptoms during the past week. A higher score means greater severity of CIPN. The maximum CIPN sensory score change (post-pre) for each patient during the intervention will be compared between the randomized treatment arms.
Changes in mean scores of pain intensity | Baseline, Week 12, and Week 24
  CIPN pain intensity will be measured using a past 7 days, 0-10 numerical rating scale diary. A higher score indicates greater pain intensity.
Changes in the total mean scores of the Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 12, and Week 24
  The PSQI is a 19-item self-reported questionnaire that assesses sleep quality for the preceding month. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Changes in the total and subscales of EORTC QLQ-C30 | Baseline, Week 12, and Week 24
  Quality of life and cancer treatment-related symptoms will be assessed using the EORTC-QLQ-C30. The QLQ-C30 consists of 30 items that are grouped within global health status/quality of life (1 - 7 points, higher scores = greater quality of life), functional (e.g., physical or cognitive; 0 - 100 transformed scores, higher = better function), or symptom (e.g., insomnia, fatigue; 0 - 100 transformed scores, higher = worse symptoms) subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Lu, MB, MPH, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu